CLINICAL TRIAL: NCT06547294
Title: Procedural and Post-Procedural Clinical Performance of a Novel Peripheral Intravenous Needle Over Catheter Device (OspreyTM)
Brief Title: Does a Novel Needle Over Catheter Device Improve First Pass Success and Decrease Complications
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Manufacturer has suspended for review
Sponsor: Community Medical Center, Toms River, NJ (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro2024001057
Record Dates: First submitted 2024-08-07; First posted 2024-08-09 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2024-08

CONDITIONS: Vascular Access Device Complications; Catheterization, Peripheral

STUDY DESIGN:
Intervention Model Description: Single arm with historical controls
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Osprey IV (Experimental): Subjects enrolled will receive the study device as part of their routine medical care.
  Interventions: Device: Osprey IV; Other: Historical Controls

INTERVENTIONS:
Device: Osprey IV — Utilization of novel needle over catheter commercial insertion device
Other: Historical Controls — Outcome rates from catheter over needle devices (traditional manner of inserting peripheral IV)

SUMMARY:
Emergency Department Patients who were to get intravenous (IV) access through routine medical care will receive it through trademarked catheter via convenience sample. Patient and clinician experience, including adverse events, will be recorded. A standardized data entry sheet will be collected at time of enrollment, and then daily thereafter while the subject has the IV. The data collected will remain anonymous.

DETAILED DESCRIPTION:
Identification of Subjects:

The emergency department is a designated participating unit providing subjects with medical care that are anticipated to be placed in the observation unit or admitted to an inpatient unit. Subjects who meet inclusion criteria will be consented to be included in the study.

Assignment of Subject Identification Number:

A unique identification number will be given to study subjects. Subject numbers will be assigned in sequential order. The subject number will consist of 6 characters. The first three characters will designate the manufacturer-specific protocol number (SVI). The last three characters will designate the subject by number in sequential order.

Informed Consent:

The nurse trained in placing this device will first consent the patient with written forms provided. All protocol nurses trained in this device will also have completed CITI training courses per our institutional guidelines.

Treatment Assignment:

Within this single arm study, subjects will be assigned to the study in a single treatment group. All patients in the convenience sample who would have received a standard stocked intravenous catheter will instead receive an Osprey catheter provided by the manufacturer. They will be compared against historical controls. Historical controls will be collected from a review of relevant literature, which has been determined to be stable across time and region.

Data Collection Method A Case Report Form (CRF) will be utilized to collect insertion related study data. The CRF will not include any patient identifying information such as name or medical identification number. The subject's demographic (age, race, and gender); baseline information (comorbidities); type of medications/fluids delivered will be documented from already captured Epic documentation.

A second Case Report Form (CRF) will be utilized to collect device performance study data. The CRF will not include any patient identifying information such as name or medical identification number. Device condition (ability to flush and obtain a blood return), Site condition (presence of redness, edema, drainage), patient response (level of pain) and dwell time will be extracted from Epic as this is the current standard practice to do so.

Active patients in the study will be maintained in a file on a secure drive that study personnel have to refer to to follow up active patients. Once active patients are no longer being followed daily, their name will be removed from that file. CRF forms will be filled out by hand and secured in a locked box. The data from both CRFs will be transcribed into a digital worksheet i.e. Microsoft Excel, which will be stored on a secured network drive maintained by the hospital.

Study Procedure Subjects will be admitted into the study according to the aforementioned criteria.

Hospital protocols will be followed for placement of the PIV. The site will be marked with date, time and initials of inserter. During and immediately after the IV placement procedure, the CRF will be initiated by staff associated with this study. If unsuccessful with first attempt at PIV placement, an attempt at another site with the same technique and device will be performed. This will be repeated according to facility policy and procedure until a successful PIV is in place or the physician decides to use an alternative therapy that no longer requires peripheral access. All catheters will be stabilized using the same form of stabilization device for uniformity in securement procedure throughout the duration of the study.

Daily assessments will occur per facility policy and procedure. An assessment will include; any level of pain and/or tenderness; presence of erythema; edema; induration; leakage of fluid or purulent drainage from the puncture site; catheter dysfunction (eg, resistance when flushing, absence of a blood return. Daily assessment will continue until the device is removed, completion of therapy or discharge. Once all the required data is collected, all de-identified data will be entered as a "data set" into the post procedure CRF for management/analysis. The final paper CRF will be placed in a study folder and maintained for record keeping and data analysis.

ELIGIBILITY:
Inclusion Criteria i. Any gender, 18 years of age or older ii. Acceptable candidate for an elective PIV as determined by physician. iii. Anticipated admission to inpatient unit.

Exclusion Criteria

1. Any gender, < 18 years old.
2. Requirement for emergent IV placement (patient's condition would be compromised if there is a delay in IV placement);
3. Previous venous grafts or surgery at the target vessel access site;
4. Currently involved in other investigational clinical trials (unless permission is granted by other study Pl)
5. Subjects who are pregnant, planning to become pregnant within 3 months of the procedure, or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Number of Attempts | 10 minutes
  The number of attempts that operator needs to access vein and secure device for proper bidirectional flow

SECONDARY OUTCOMES:
Blood culture contamination rates | 1 week
  Proportion of blood culture specimens (when drawn) that are reported with contaminants
Flushing characteristic | 10 minutes
  whether operator finds flow into patient to be impeded or unimpeded
Patient discomfort | 10 minutes
  Patient's self assessment of level of pain experienced by insertion
Time to removal | 1 week
  Total days device remained in place
Removal reason | 1 week
  If removed for device failure vs cessation of therapy
Edema | 1 week
  Presence of edema
Redness | 1 week
  Presence of redness
Drainage | 1 week
  Presence of drainage
Site Pain | 1 week
  Presence of site pain

CONTACTS AND LOCATIONS:
Overall Officials: Gerado Chiricolo, MD, Principal Investigator — Robert Wood Johnson Barnabas Health
Locations (1):
- Robert Wood Johnson Barnabas Health Community Medical Center, Toms River, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Device White Paper — https://www.skydancevascular.com/wp-content/uploads/2022/05/White-Paper-Advancing-Toward-the-Expansion-of-Catheter-Related-Blood-Stream-Infection-Reporting-to-Include-PIVs.pdf